CLINICAL TRIAL: NCT03572777
Title: A Randomized Controlled Study: Concomitant Versus Hybrid Therapy in the Treatment of Helicobacter Pylori Infection
Brief Title: Comparison of Therapy in Treatment of Patients With Helicobacter Pylori Infection: Concomitant Versus Hybrid Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Mestrovic (Other)
Collaborators: University Hospital of Split (Other); University of Split, School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Antonio Mestrovic, Sponsor-Investigator, University of Split, School of Medicine
Organization: University of Split, School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003-08/18-03/0001
Record Dates: First submitted 2018-05-24; First posted 2018-06-28 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori, eradication, hybrid therapy, concomitant therapy
MeSH Terms: interventions — Hybrid Renal Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concomitant therapy (Active Comparator): Amoxicillin ('Amoksicilin') 1 g bid, metronidazole ('Medazol')500 mg bid, clarithromycin ('Makcin')500 mg bid and esomeprazole ('Emanera')40 mg bid for 14 days.
  Interventions: Drug: Concomitant therapy
- Hybrid therapy (Active Comparator): Amoxicillin ('Amoksicilin') 1 g bid and esomeprazole ('Emanera') 40 mg bid for 14 days, with metronidazole ('Medazol')500 bid and clarithromycin ('Makcin') 500 mg bid for the last 7 days.
  Interventions: Drug: Hybrid therapy

INTERVENTIONS:
Drug: Concomitant therapy — Amoxicillin ('Amoksicilin') 1 g bid 14 days.
  Arms: Concomitant therapy
Drug: Concomitant therapy — Clarithromycin ('Makcin') 500 mg bid for 14 days
  Arms: Concomitant therapy
Drug: Concomitant therapy — Metronidazole ('Medazol') 500 mg bid for 14 days
  Arms: Concomitant therapy
Drug: Concomitant therapy — Esomeprazole ('Emanera') 40 mg bid for 14 days
  Arms: Concomitant therapy
Drug: Hybrid therapy — Amoxicillin ('Amoksicilin') 1 g bid 14 days
  Arms: Hybrid therapy
Drug: Hybrid therapy — Esomeprazole ('Emanera') 40 mg bid for 14 days
  Arms: Hybrid therapy
Drug: Hybrid therapy — Clarithromycin ('Makcin') 500 mg bid for the last 7 days
  Arms: Hybrid therapy
Drug: Hybrid therapy — Metronidazole ('Medazol') 500 mg bid for the last 7 days
  Arms: Hybrid therapy

SUMMARY:
The aim of the study is to compare the effectiveness of two therapeutic protocols in the treatment of Helicobacter pylori infection.

The hypothesis of our research is that the two therapeutic options (hybrid and concomitant therapy) will be equally successful in the treatment of Helicobacter pylori infection. In other words, in both therapeutic groups we expect successful treatment of Helicobacter pylori infection in or more than 90 % of patients.

In other studies, both therapeutic options have the same efficacy in treating H. pylori infection. On the other had there are no studies available in Croatia to compare the effectiveness of these therapeutic options so far, which is the main objective of our research. The secondary goals of our study will be: the existence of differences in the occurrence of possible side effects, as well as the compliance between patients in both therapeutic options. It is also our aim to compare the quality of life of patients with Helicobacter pylori infection before and after treatment, via a questionnaire that is common for this purpose.

The study is expected to include a total of 120 patients (60 patients in each therapy group), and the planned duration is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infection (documented by: positive antigen stool test, or positive urease rapid test obtained during upper endoscopy, or Helicobacter pylori in histological finding, or positive C-urea breath test; according to recent Maastricht V guidelines;
* written informed consent

Exclusion Criteria:

* age under 18
* previously treatment of Helicobacter pylori infection
* malignancy of stomach or other site
* history of taking proton pump inhibitors, H2 antagonist, bismuth or antibiotics (amoxicillin, metronidazole, clarithromycin) in previous month
* significant underlying disease (renal failure, psychiatric disorders)
* history of allergic reactions to any medications used in study
* refuse to participate in study
* breastfeeding and pregnancy
* quitting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori status one month after treatment. | One month after finishing with therapy.
  Helicobacter pylori status (positive or negative), will be measured by stool test, one month after finishing with therapy.

SECONDARY OUTCOMES:
Compliance of patients in both therapy groups in treatment of Helicobacter pylori infection. | One month after finishing with therapy.
  Compliance will be measured by counting pills that were taken during therapy. More than or equal 80 % of taken pills will be consider as good compliance
Adverse effects of therapy in both groups in treatment of Helicobacter pylori infection. | One month after finishing with therapy.
  Patients will be ask to report any adverse effect occured during treatment. They will be divided in groups according to degree of limiting daily activities: no adverse effects; mild (no limit of activities); moderate (partially limited activities); severe (completely limited activities).

OTHER OUTCOMES:
Quality of life before and after eradication therapy | One month after therapy
  Quality of life before and after eradication (both groups combined) therapy will be reported by The Gastrointestinal Symptom Rating Scale (GSRS) questionnaire. GSRS questionnaire: 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents no discomfort at all, 2 - minor discomfort, 3 -mild discomfort, 4 - moderate discomfort, 5 -moderately severe discomfort, 6 -severe discomfort, 7 - very severe discomfort
Quality of life before and after eradication therapy between hybrid and concomitant group. | One month after therapy
  Quality of life before and after eradication therapy will be reported by the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire comparing both groups. GSRS questionnaire: 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents no discomfort at all, 2 - minor discomfort, 3 -mild discomfort, 4 - moderate discomfort, 5 -moderately severe discomfort, 6 -severe discomfort, 7 - very severe discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Meštrović, MD, Principal Investigator — University Hospital Centre Split, Croatia
Locations (1):
- University Hospital Centre Split, Split, Croatia

REFERENCES:
- [Derived] Mestrovic A, Perkovic N, Bozic J, Pavicic Ivelja M, Vukovic J, Kardum G, Puljiz Z, Tonkic A. Randomised clinical trial comparing concomitant and hybrid therapy for eradication of Helicobacter pylori infection. PLoS One. 2020 Dec 30;15(12):e0244500. doi: 10.1371/journal.pone.0244500. eCollection 2020. PMID 33378403